CLINICAL TRIAL: NCT06361394
Title: The Impacts of Mindfulness on Psychological Wellbeing and Nursing Competencies Among Nursing Students: a Longitudinal Study of Mindfulness Education Course Design, Implementation, and Effectiveness Verification
Brief Title: The Impacts of Mindfulness on Psychological Wellbeing Among Nursing Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University of Science and Technology (Other)
Responsible Party: Principal Investigator, Ya-Chu Hsiao, professor, Chang Gung University of Science and Technology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CORPFIN0021
Record Dates: First submitted 2024-02-15; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Students
Keywords: Mindfulness; Empathy; Stress; Anxiety; Competency
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The experimental group will enroll in the elective course named "Mindfulness and Happiness," which will consist of 2 hours every week for a continuous period of 18 weeks. The comparison group will not participate in this course.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- receive a new elective course (Experimental): The experimental group will enroll in the elective course named "Mindfulness and Happiness," which will consist of 2 hours every week for a continuous period of 18 weeks.
  Interventions: Other: mindfulness course
- not receive a new elective course (No Intervention): The comparison group do not enroll in the new elective course named "Mindfulness and Happiness,"

INTERVENTIONS:
Other: mindfulness course — The experimental group will enroll in the elective course named "Mindfulness and Happiness," which will consist of 2 hours every week for a continuous period of 18 weeks. The comparison group will not participate in this course.
  Arms: receive a new elective course

SUMMARY:
The aims of this study are to develop a mindfulness-based course for nursing students. As well as, to verify the effects on psychological well-being (mindfulness, stress, and anxiety) and nursing professional related competences (empathy, clinical practicum stress, nursing competency) among nursing students.

DETAILED DESCRIPTION:
A quasi-experimental study design will be used to examine the effects of a new elective course. Convenient sampling will be used to invite nursing students at a university of science and technology in Taiwan. The data will be collected four seven times, including baseline (T0), the end of the course (T1), before and after the nursing practicum (T2, T3).

Participants who enroll in an elective course in mindfulness education constitute the experimental group, while those who do not enroll in the elective form the comparison group. The total number of participants will be 240. Participants will be excluded if they are unwilling to participate in the study or do not complete the consent form.

Intervention: The experimental group will enroll in the elective course named "Mindfulness and Happiness," which will consist of 2 hours every week for a continuous period of 18 weeks. The comparison group will not participate in this course. The elective course is designed using the ADDIE model (Analysis, Design, Development, Implementation, Evaluation) and is based on Mindfulness-based Stress Reduction principles.

ELIGIBILITY:
Inclusion Criteria:

* Nursing students who participated in the elective mindfulness course

Exclusion Criteria:

* under 18 years

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-07-25 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
perceived stress at baseline | Data were collected before course intervention
  The Cohen's Perceived stress scale is a validated multidimensional measure that assesses individuals' stress level. Higher score indicated higher level of stress.
perceived stress at T0 | Data were collected end the course intervention, around 5 months after baseline data collection.
  The Cohen's Perceived stress scale is a validated multidimensional measure that assesses individuals' stress level. Higher score indicated higher level of stress.
perceived stress at T1 | Data were collected before the nursing practicum, around 6 months after baseline data collection.
  The Cohen's Perceived stress scale is a validated multidimensional measure that assesses individuals' stress level. Higher score indicated higher level of stress.
perceived stress at T2 | Data were collected after the nursing practicum,around 7 months after baseline data collection.
  The Cohen's Perceived stress scale is a validated multidimensional measure that assesses individuals' stress level. Higher score indicated higher level of stress.
anxiety disorder at baseline | Data were collected before course intervention
  Löwe's the Generalized Anxiety Disorder 7-Item Scale(GAD-7) generalized anxiety disorder 7-item scale is a validated measure that assesses individuals' anxiety level. higher score indicated higher level of anxiety.
anxiety disorder at T0 | Data were collected end course intervention,around 5 months after baseline data collection.
  Löwe's the Generalized Anxiety Disorder 7-Item Scale(GAD-7) generalized anxiety disorder 7-item scale is a validated measure that assesses individuals' anxiety level. higher score indicated higher level of anxiety.
anxiety disorder at T1 | Data were collected before the nursing practicum,around 6 months after baseline data collection.
  Löwe's the Generalized Anxiety Disorder 7-Item Scale(GAD-7) generalized anxiety disorder 7-item scale is a validated measure that assesses individuals' anxiety level. higher score indicated higher level of anxiety.
anxiety disorder at T2 | Data were collected after the nursing practicum, around 7 months after baseline data collection.
  Löwe's the Generalized Anxiety Disorder 7-Item Scale(GAD-7) generalized anxiety disorder 7-item scale is a validated measure that assesses individuals' anxiety level. higher score indicated higher level of anxiety.
mindful attention awareness at baseline | Data were collected before course intervention
  Brown & Ryan's Mindful Attention Awareness Scale is a validated multidimensional measure that assesses individuals' mindful quality.higher score indicated higher level mindfulness.
mindful attention awareness at T0 | Data were collected end the course intervention, around 5 months after baseline data collection.
  Brown & Ryan's Mindful Attention Awareness Scale is a validated multidimensional measure that assesses individuals' mindful quality.higher score indicated higher level mindfulness.
mindful attention awareness at T1 | Data were collected before the nursing practicum,around 6 months after baseline data collection.
  Brown & Ryan's Mindful Attention Awareness Scale is a validated multidimensional measure that assesses individuals' mindful quality.higher score indicated higher level mindfulness.
mindful attention awareness at T2 | Data were collected after the nursing practicum.around 7 months after baseline data collection.
  Brown & Ryan's Mindful Attention Awareness Scale is a validated multidimensional measure that assesses individuals' mindful quality.higher score indicated higher level mindfulness.
empathy at baseline | Data were collected before the course intervention
  Jefferson scale of empathy Chinese version is a validated multidimensional measure that assesses individuals' empathy level.higher score indicated higher level empathy.
empathy at at T0 | Data were collected end the course intervention, around 5 months after baseline data collection.
  Jefferson scale of empathy Chinese version is a validated multidimensional measure that assesses individuals' empathy level.higher score indicated higher level empathy.
empathy at at T1 | Data were collected before the nursing practicum,around 6 months after baseline data collection.
  Jefferson scale of empathy Chinese version is a validated multidimensional measure that assesses individuals' empathy level.higher score indicated higher level empathy.
empathy at at T2 | Data were collected after the nursing practicum.around 7 months after baseline data collection.
  Jefferson scale of empathy Chinese version is a validated multidimensional measure that assesses individuals' empathy level. higher score indicated higher level empathy.
practicum stress at T1 | Data were collected before the nursing practicum, around 6 months after baseline data collection.
  The perceived practicum stress scale is a validated multidimensional measure that assesses individuals' nursing stress from practicum.higher score indicated higher level stress of practicum.
practicum stress at T2 | Data were collected after the nursing practicum,around 7 months after baseline data collection.
  The perceived practicum stress scale is a validated multidimensional measure that assesses individuals' nursing stress from practicum.higher score indicated higher level stress of practicum.
Nursing Competence at T1 | Data were collected before the nursing practicum,around 6 months after baseline data collection.
  The Competence Scale for Clinical Nurse (CSCN) is a validated multidimensional measure that assesses nursing student' nursing competence. higher score indicated higher level of nursing competence.
Nursing Competence at T2 | Data were collected after the nursing practicum,around 7 months after baseline data collection.
  The Competence Scale for Clinical Nurse (CSCN) is a validated multidimensional measure that assesses nursing student' nursing competence. higher score indicated higher level of nursing competence.

CONTACTS AND LOCATIONS:
Locations (1):
- Ya-Chu Hsiao, Taoyuan, N/A = Not Applicable, Taiwan

IPD SHARING:
Plan to Share IPD: No
IRB does not allow